CLINICAL TRIAL: NCT00163436
Title: Comparison of the Efficacy and Safety of 160 mcg Ciclesonide Administered Once Daily in the Evening With or Without Different Spacer Types in Patients With Asthma
Brief Title: Efficacy and Safety of Ciclesonide Administered With or Without Different Spacers in Patients With Asthma (12 to 75 y) (BY9010/M1-145)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BY9010/M1-145
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the present study is to investigate the efficacy and safety of ciclesonide on lung function and safety. Ciclesonide will be inhaled at one dose level once daily, using an inhaler device with or without spacer. The study duration consists of a baseline period (1 to 3 weeks) and a treatment period (12 weeks).

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* History of persistent bronchial asthma for at least 6 months
* Good health with the exception of asthma

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* Smoking history with ≥10 cigarette pack years
* Pregnancy
* Intention to become pregnant
* Breast feeding
* Lack of safe contraception
* Previous enrolment into the current study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2005-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
FEV1.

SECONDARY OUTCOMES:
FVC
morning and evening PEF from diaries
asthma symptom score
use of rescue medication
number of patients with an asthma exacerbation
time to the first asthma exacerbation
percentage of days on which patient perceived asthma control
percentage of nocturnal awakening-free days
percentage of rescue medication-free days
percentage of asthma symptom-free days
adverse events
physical examination
vital signs
standard laboratory work-up
8 am serum cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (61):
- Canada (15):
  - Altana Pharma/Nycomed, La Malbaie, Quebec
  - Altana Pharma/Nycomed, London
  - Altana Pharma/Nycomed, London,ON
  - Altana Pharma/Nycomed, Mississauga
  - Altana Pharma/Nycomed, Montreal, Quebec
  - Altana Pharma/Nycomed, Québec
  - Altana Pharma/Nycomed, Richmond Hill
  - Altana Pharma/Nycomed, Sainte-Foy, Quebec
  - Altana Pharma/Nycomed, Saskatoon,SK
  - Altana Pharma/Nycomed, Scarborough,ON
  - Altana Pharma/Nycomed, Toronto
  - Altana Pharma/Nycomed, Vancouver, BC
  - Altana Pharma/Nycomed, Winnipeg
  - Altana Pharma/Nycomed, Winnipeg MB
  - Altana Pharma/Nycomed, Woodstock
- France (15):
  - Altana Pharma/Nycomed, Aix-en-Provence
  - Altana Pharma/Nycomed, Chauny
  - Altana Pharma/Nycomed, Ferolles-Attily
  - Altana Pharma/Nycomed, Grasse
  - Altana Pharma/Nycomed, La Rochelle
  - Altana Pharma/Nycomed, La Teste-de-Buch
  - Altana Pharma/Nycomed, Libourne
  - Altana Pharma/Nycomed, Lille
  - Altana Pharma/Nycomed, Martigues
  - Altana Pharma/Nycomed, Montbrison
  - Altana Pharma/Nycomed, Montpellier
  - Altana Pharma/Nycomed, Nice
  - Altana Pharma/Nycomed, Nîmes
  - Altana Pharma/Nycomed, Saint-Laurent-du-Var
  - Altana Pharma/Nycomed, Saint-Quentin
- Germany (5):
  - Altana Pharma/Nycomed, Berlin
  - Altana Pharma/Nycomed, Oschersleben
  - Altana Pharma/Nycomed, Rüdersdorf
  - Altana Pharma/Nycomed, Schwetzingen
  - Altana Pharma/Nycomed, Weinheim
- Hungary (12):
  - Altana Pharma/Nycomed, Balassagyarmat
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Budapet
  - Altana Pharma/Nycomed, Érd
  - Altana Pharma/Nycomed, Gyula
  - Altana Pharma/Nycomed, Komárom
  - Altana Pharma/Nycomed, Miskolc
  - Altana Pharma/Nycomed, Mosdós
  - Altana Pharma/Nycomed, Nyiregyháza
  - Altana Pharma/Nycomed, Pécs
  - Altana Pharma/Nycomed, Szeged
  - Altana Pharma/Nycomed, Székesfehérvár
- India (9):
  - Altana Pharma/Nycomed, Bangalore
  - Altana Pharma/Nycomed, Chennai
  - Altana Pharma/Nycomed, Coimbatore
  - Altana Pharma/Nycomed, Coimbatore, Tamilnadu
  - Altana Pharma/Nycomed, Goa
  - Altana Pharma/Nycomed, Kalaburagi
  - Altana Pharma/Nycomed, Mumbai
  - Altana Pharma/Nycomed, Mumbai, Dadar (E)
  - Altana Pharma/Nycomed, Pune
- Italy (5):
  - Altana Pharma/Nycomed, Florence
  - Altana Pharma/Nycomed, Milan
  - Altana Pharma/Nycomed, Napoli
  - Altana Pharma/Nycomed, Pordenone
  - Altana Pharma/Nycomed, Verona

REFERENCES:
- See also: BY9010-MI-145-RDS-2007-05-21.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4524&filename=BY9010-MI-145-RDS-2007-05-21.pdf